CLINICAL TRIAL: NCT07069166
Title: Evaluation of Para-Probiotic Toothpaste and Mouthwash on Periodontal Health and Glycemic Control in Diabetic Patients: A Randomized Controlled Trial
Brief Title: Para-Probiotic Oral Care in Periodontal Patients With Type 2 Diabetes
Acronym: PPDM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-PPDM2
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis; Type 2 Diabetes Mellitus (T2DM)
Keywords: Para-probiotics; Periodontitis; Type 2 Diabetes Mellitus; Biorepair; Oral microbiota; Glycated hemoglobin (HbA1c); Chlorhexidine; Non-surgical periodontal therapy; Randomized controlled trial
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Para-Probiotic Oral Care Group (Experimental): Participants receive standard non-surgical periodontal therapy and use para-probiotic toothpaste (Biorepair Plus Parodontogel) and para-probiotic mouthwash (Biorepair Plus), twice daily for 15 days after each recall visit, over a 6-month period.
  Interventions: Drug: Para-probiotic oral care
- Chlorhexidine Oral Care Group (Active Comparator): Participants receive standard non-surgical periodontal therapy and use toothpaste and mouthwash containing 0.20% chlorhexidine, twice daily for 15 days after each recall visit, over a 6-month period.
  Interventions: Drug: Chlorhexidine oral care

INTERVENTIONS:
Drug: Para-probiotic oral care — This intervention includes the home use of a para-probiotic-based toothpaste (Biorepair Plus Parodontogel) and mouthwash (Biorepair Plus with para-probiotics), applied twice daily for 15 days after each recall visit, over a 6-month period. The products contain microRepair® (zinc hydroxyapatite), lactoferrin, zinc PCA, and para-probiotic extracts aimed at modulating the oral microbiota and improving periodontal health.
  Arms: Para-Probiotic Oral Care Group
Drug: Chlorhexidine oral care — This intervention includes the home use of toothpaste and mouthwash containing 0.20% chlorhexidine digluconate, applied twice daily for 15 days after each recall visit, over a 6-month period. Chlorhexidine is used for its antimicrobial properties to control dental plaque and gingival inflammation.
  Arms: Chlorhexidine Oral Care Group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of a para-probiotic-based oral care protocol in improving periodontal health and glycemic control in patients with type 2 diabetes mellitus (T2DM).

A total of 40 adult patients (aged 18-70) with diagnosed periodontitis and T2DM will be enrolled and randomly assigned to two treatment groups. Both groups will receive standard non-surgical periodontal therapy. The test group will use para-probiotic toothpaste and mouthwash (Biorepair Plus Parodontogel and Biorepair Plus mouthwash) twice daily for 15 days after each recall visit, while the control group will use toothpaste and mouthwash containing 0.20% chlorhexidine on the same schedule.

Clinical evaluations will be conducted at baseline (T0), 3 months (T1), and 6 months (T2), assessing key periodontal parameters including clinical attachment level (CAL), bleeding on probing (BoP), probing pocket depth (PPD), plaque index (PI), and glycemic control via hemoglobin A1c (HbA1c) levels. Patient satisfaction with treatment will be assessed using a questionnaire at T1 and T2.

The primary objective is to evaluate the change in CAL from baseline to 6 months. Secondary objectives include the evaluation of changes in BoP, PPD, PI, HbA1c, and patient-reported satisfaction.

This study seeks to determine whether para-probiotic oral care products can offer clinical benefits for periodontal disease management and systemic glycemic control in diabetic patients, potentially serving as a natural adjunct to conventional periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Diagnosis of periodontitis (Stage II or III; Grade B or C)
* Presence of at least one periodontal pocket per side of the mouth, with a maximum of 20 teeth presenting pathological probing depths
* Presence of both single- and multi-rooted teeth
* Type 2 diabetes mellitus diagnosed at least one year prior to enrollment
* Good general health status and ability to comply with study protocol
* Written informed consent provided

Exclusion Criteria:

* Presence of cardiac pacemakers
* History of neurological disorders
* History of psychiatric disorders
* Current pregnancy or breastfeeding
* Steroid-induced diabetes mellitus
* Inability or unwillingness to attend follow-up visits or adhere to home oral care instructions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in mean Clinical Attachment Level (CAL) | Baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2)
  This outcome measures the difference in mean Clinical Attachment Level (CAL) between baseline and the 6-month follow-up in patients with periodontitis and type 2 diabetes mellitus, randomized to receive either para-probiotic-based or chlorhexidine-based oral care after standard non-surgical periodontal therapy. CAL will be assessed in millimeters at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) using a calibrated manual periodontal probe. Measurements will be performed at three predefined timepoints: at baseline (T0, Day 0) before the start of treatment; at three months (T1, approximately Day 90) as an intermediate evaluation; and at six months (T2, approximately Day 180), which represents the final endpoint. The primary endpoint is defined as the difference in mean CAL per patient between the baseline and the 6-month follow-up.

SECONDARY OUTCOMES:
Change in Bleeding on Probing (BoP) score | Baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2)
  This outcome measures the variation in Bleeding on Probing (BoP) between baseline and follow-up visits in patients receiving either para-probiotic or chlorhexidine oral care. BoP is assessed using a calibrated periodontal probe inserted into the gingival sulcus at six sites per tooth. A site is considered positive if bleeding occurs within 15 seconds of probing. The BoP score is expressed as the percentage of bleeding sites out of the total number of sites examined for each patient. Higher scores indicate a greater degree of gingival inflammation. Measurements will be recorded at baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2). The endpoint is defined as the change in mean BoP score between T0 and T2.
Change in Probing Pocket Depth (PPD) score | Baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2)
  This outcome assesses the variation in Probing Pocket Depth (PPD) between baseline and follow-up visits in patients receiving either para-probiotic or chlorhexidine oral care. PPD is measured in millimeters using a calibrated UNC-15 periodontal probe inserted into the gingival sulcus at six sites per tooth. The depth is recorded as the distance from the gingival margin to the bottom of the periodontal pocket. The PPD score is calculated as the mean depth of all recorded sites per patient. Higher values indicate more severe periodontal involvement. Measurements will be taken at baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2). The endpoint is defined as the change in mean PPD score between T0 and T2.
Change in Plaque Index (PI) score | Baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2)
  This outcome evaluates the variation in the Plaque Index (PI) score between baseline and follow-up in both study groups. PI is determined by visually assessing the presence of dental plaque on four surfaces per tooth (distal, mesial, buccal, and lingual/palatal) after disclosing agent application. The score is expressed as the percentage of plaque-positive sites over the total number of examined sites per patient. Higher scores indicate poorer oral hygiene and greater plaque accumulation. Measurements are collected at baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2). The endpoint is the change in mean PI score between T0 and T2.
Change in glycated hemoglobin (HbA1c) level | Baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2)
  This outcome measures the variation in glycated hemoglobin (HbA1c) levels between baseline and follow-up in patients undergoing para-probiotic or chlorhexidine oral care. HbA1c is measured using standardized blood assays and reflects average blood glucose control over the previous 8-12 weeks. The value is expressed as a percentage of total hemoglobin. Lower values indicate better glycemic control. Measurements are performed at baseline (T0), 3-month follow-up (T1), and 6-month follow-up (T2). The endpoint is the change in mean HbA1c level between T0 and T2.
Change in patient satisfaction score | 3-month follow-up (T1) and 6-month follow-up (T2)
  This outcome evaluates the variation in patient-reported satisfaction with the oral care protocol. Satisfaction is assessed using a structured, self-administered questionnaire consisting of Likert-scale items (ranging from 1 = very dissatisfied to 5 = very satisfied) regarding taste, ease of use, perceived effectiveness, and overall comfort. The total score is calculated as the mean of all items per patient. Higher scores reflect greater satisfaction. The questionnaire is administered at 3-month follow-up (T1) and 6-month follow-up (T2). The endpoint is the change in mean satisfaction score between T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.